CLINICAL TRIAL: NCT03220152
Title: Implementation of the Pre-Exposure Prophylaxis (PrEP) to HIV in Brazilian Transgender Women
Brief Title: Implementation of PrEP to HIV in Brazilian Transgender Women
Acronym: PrEParadas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oswaldo Cruz Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrEParadas
Record Dates: First submitted 2017-07-06; First posted 2017-07-18 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: HIV, Prevention
MeSH Terms: interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- emtricitabine / tenofovir 200/300 mg (Experimental): emtricitabine / tenofovir 200/300 mg Fixed dose combination of emtricitabine / tenofovir 200/300 mg once daily orally during one year.
  Interventions: Drug: emtricitabine / tenofovir 200/300 mg

INTERVENTIONS:
Drug: emtricitabine / tenofovir 200/300 mg — Fixed dose combination of emtricitabine / tenofovir 200/300 mg once daily orally during one year
  Other Names: Truvada

SUMMARY:
Subjects preliminarily eligible who choose to receive PrEP will be included after obtaining the informed consent and confirmation of eligibility within 45 days after the screening visit.

Once included, participants will be examined in a follow-up visit performed four weeks later and evaluated for evidence of seroconversion to HIV, medication compliance and clinical toxicity. The second follow-up visit will occur at 12th week and every 12 weeks successively (quarterly). Quarterly visits include HIV testing, serum creatinine and counseling on medication compliance and risk reduction.

The study has a total of 6 visits plus 2 extra visits for those participants enrolled in the PK study. In all visits will be assessed the risks, HIV testing will be performed, monitoring of renal function and dispensing of the drug Truvada [emtricitabine 1 tablet (FTC) / tenofovir (TDF) (200/300 mg) once a day orally for 12 months].

Participants who have completed 48 weeks of follow-up or prematurely discontinue a PrEP will be encouraged to return for a follow-up visit after discontinuation of medication for monitoring of the status and evaluation of HIV as the resolution of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Male (at birth) AND transgender women identity;
* Willing and able to provide informed consent in writing;
* Age = or > 18 years;
* Not infected by HIV-1, in accordance with the flowchart of testing from Brazilian Ministry of Health;
* Evidence risk for acquiring HIV-1, including any of the following:
* Anal or vaginal sex without a condom with two or more men or transgender women in the last 12 months, or
* 2 or more episodes of anal sex with at least one HIV+ sexual partner HIV + in the last 12 months, or
* Sex with a man or trans woman and diagnosis or report of any of the following STDs in the last 12 months: syphilis, rectal gonorrhea or chlamydial infection in the rectum.;
* Report of exchanging sex for money, presents, shelter or drugs.
* Able to provide a residential address or contact phone itself, or two personal contacts who would know about his whereabouts during the study period demonstrative;
* Adequate renal function: Creatinine clearance > or = 60 ml / min, estimated by the formula modification of diet in renal disease (MDRD, from English 'Modification of Diet in Renal Disease') within 45 days of enrollment;
* urine Tape with negative result or showing only traces of protein within 45 days prior to enrollment;

Exclusion Criteria:

* Signs or symptoms of acute HIV infection,which is confirmed by laboratory examination in subsequent samples;
* Active and severe infections previously diagnosed, including active tuberculosis or osteomyelitis and all infections requiring parenteral antibiotics (except STD that require intramuscular injections of antibiotics);
* clinically significant active medical problems, including heart disease poorly controlled (eg, symptoms ischemia, congestive heart failure) previously diagnosed malignancy, or which will require additional treatment;
* Patients with positive tests for antigens of hepatitis B surface (HBsAg);
* History of pathological bone fractures unrelated to trauma;
* Patients using any of the following: ARV, including nucleoside inhibitors, non-nucleoside reverse transcriptase inhibitors, protease inhibitors and antiretroviral agents under study, treatment with interferon (alpha, beta, or gamma) or interleukin (e.g. ,IL-2), with potential significant nephrotoxic agents, other agents which may inhibit or compete for renal elimination via active tubular secretion (eg probenecid) and / or other agents under study;
* Participation in a clinical trial using concomitant agents under investigation, including placebo-controlled trials using such agents;
* Patients who have any condition at the time of inclusion in the study, according to the opinion of the investigator, may prevent the provision of informed consent, make study participation unsafe, complicate data interpretation, or interfere anyway with the achievement of project objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male (at birth) AND transgender women identity;
Enrollment: 120 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Compliance to study treatment | 2 years
  Number of volunteers who keep the study treatment during 24 months Correlation of socio-demographic factors of acceptance and refusal Duration of PrEP Side effects and toxicities, including elevations of creatinine Adherence to PrEP: number of tablets per day, patterns of adherence Number of male sexual partners, by serostatus and condom use, and episodes of anal sex by partner serostatus, the interviewee practices and condom use.

SECONDARY OUTCOMES:
HIV seroconversions rate | 2 years
  Number of patients who become HIV-infected
Maximum Plasma Concentration [Cmax] of FTC / TDF | 2 years
  Compare FTC/TDF Cmax between volunteers using or not hormones
Area Under the Curve [AUC] of FTC / TDF | 2 years
  Compare FTC/TDF AUC between volunteers using or not hormones

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Infectologia Evandro Chagas (INI) - Fiocruz, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cattani VB, Jalil EM, Eksterman L, Torres T, Wagner Cardoso S, Castro CRV, Monteiro L, Wilson E, Bushman L, Anderson P, Veloso VG, Grinsztejn B, Estrela R; PrEParadas study team. Estradiol and Spironolactone Plasma Pharmacokinetics Among Brazilian Transgender Women Using HIV Pre-Exposure Prophylaxis: Analysis of Potential Interactions. Clin Pharmacokinet. 2023 Jul;62(7):1031-1041. doi: 10.1007/s40262-023-01248-0. Epub 2023 Jun 1. PMID 37261664
- [Derived] Jalil EM, Torres TS, Luz PM, Monteiro L, Moreira RI, de Castro CRV, Leite IDC, Cunha M, de Cassia Elias Estrela R, Ramos M, Hoagland B, Wagner Cardoso S, Anderson P, Veloso VG, Wilson E, Grinsztejn B; PrEParadas Study Team. Low PrEP adherence despite high retention among transgender women in Brazil: the PrEParadas study. J Int AIDS Soc. 2022 Mar;25(3):e25896. doi: 10.1002/jia2.25896. PMID 35255199